CLINICAL TRIAL: NCT03763227
Title: Efficacy and Safety of Intravitreal Ranibizumab (Lucentis®) Injection in the Treatment of Non-leaking Macular Cysts in Patients With Retinal Dystrophy.
Brief Title: Intravitreal Ranibizumab (Lucentis®) in the Treatment of Non-leaking Macular Cysts in Retinal Dystrophy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sultan Qaboos University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MREC 883
Record Dates: First submitted 2018-12-01; First posted 2018-12-04 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Retinal Dystrophies
MeSH Terms: conditions — Retinal Dystrophies | interventions — Injections; Carbonic Anhydrase Inhibitors; carboxyamido-triazole; Therapeutics

STUDY DESIGN:
Intervention Model Description: Phase 1: Patients with best corrected visual acuity (BCVA) < 0.5 will receive carbonic anhydrase inhibitors (CAI) [oral acetazolamide 500mg/day or topical brinzolamide twice daily] and followed up for three months. Phase 2: Patients who do not show an adequate response with CAI will receive three 0.5mg IVR injection at monthly intervals.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Carbonic Anhydrase Inhibitor (CAI) Arm (Active Comparator): Patients who have received carbonic anhydrase inhibitor (CAI) therapy namely oral acetazolamide or topical brinzolamide
  Interventions: Drug: Carbonic Anhydrase Inhibitor (CAI) therapy
- Intravitreal ranibizumab (IVR) arm (Experimental): Intravitreal ranibizumab (IVR) injection administered to patients who have not shown adequate response or who have not tolerated CAI therapy
  IVR therapy = Three 0.5mg IVR injection at monthly intervals
  Interventions: Drug: Intravitreal ranibizumab (IVR) injection

INTERVENTIONS:
Drug: Intravitreal ranibizumab (IVR) injection — Intravitreal ranibizumab (IVR) injection in patients with retinal dystrophy and macular cysts who have not responded to treatment with carbonic anhydrase inhibitors
  Arms: Intravitreal ranibizumab (IVR) arm
Drug: Carbonic Anhydrase Inhibitor (CAI) therapy — Carbonic anhydrase therapy (Oral or Topical) in patients with retinal dystrophy and macular cysts
  Other Names: CAI
  Arms: Carbonic Anhydrase Inhibitor (CAI) Arm

SUMMARY:
To evaluate the efficacy and safety of intravitreal ranibizumab (IVR) injection in the treatment of non-leaking macular cysts in patients with retinal dystrophy.

Material and Methods:

Design - Prospective, nonrandomized, nonblinded, clinical trial. Participants - Patients >18 years diagnosed with retinal dystrophies and non-leaking macular cysts between Jan 2015 and July 2018 in 1 center.

Methods - Phase 1: Patients with best corrected visual acuity (BCVA) < 0.5 will receive carbonic anhydrase inhibitors (CAI) [oral acetazolamide 500mg/day or topical brinzolamide twice daily] and followed up for three months. Phase 2: Patients who do not show an adequate response with CAI will receive three 0.5mg IVR injection at monthly intervals.

Outcome - 1) Significant reduction (> 10%) of the central macular thickness (CMT), 2) Improvement (> 1 line) in BCVA 3) Presence of any complication.

DETAILED DESCRIPTION:
The treatment of cystoid macular edema (CME) in retinitis pigmentosa (RP) is well established in medical literature. These treatments include topical and oral carbonic anhydrase inhibitors (CAI), intravitreal triamcinolone acetonide, and laser photocoagulation. Oral acetazolamide, a carbonic anhydrase inhibitor (CAI), was found to be effective in the treatment of RP related CME with improvement in both visual acuity and fundus fluorescein angiography (FFA). However, some patients may not benefit from the treatment, or do not tolerate it, while others may develop rebound CME with prolonged use of at least 8 to 12 weeks.

An emerging treatment modality for CME in RP is the use of intravitreal injections of anti-vascular endothelial growth factors (anti-VEGF) such as bevacizumab (Avastin®) and ranibizumab (Lucentis®). Anti-VEGF has been used successfully for treating diabetic macular edema, and macular edema secondary to retinal vein occlusion and choroidal neovascularization, with limited side effects.

A subset of patients with retinal dystrophy develop non-leaking macular cysts that can be confused with CME on ophthalmoscopy and optical coherence tomography (OCT). FFA establishes the cavitary nature of the maculopathy, with no hyperfluorescence seen on angiography compared with leakage seen in patients with CME and retinal dystrophy.

CAI may promote resolution of the non-leaking macular cysts. There are limited studies that explore the effect of anti-VEGF specifically on non-leaking macular cysts in retinal dystrophies.

Aims:

- Assess the efficacy of intravitreal ranibizumab (IVR) injection in the treatment of non-leaking macular cystic lesions in patients with retinal dystrophy that have not responded to therapy with oral or topical CAI.

Objectives:

* Delineate the entity of non-leaking macular cysts by OCT and FFA.
* Assess the efficacy of short-term oral and topical CAI treatment on non-leaking macular cysts in retinal dystrophies.
* Study the visual response and structural resolution of non-leaking macular cysts in response to IVR.

Design: Two-phase prospective, non-randomized, open-label, comparative interventional, clinical trial.

Inclusion criteria:

1. Omani patients over 18 years old
2. Retinal dystrophy and non-leaking macular cysts confirmed by fundus examination, electroretinography (ERG), OCT, FFA and genetic testing.
3. Capacity and cooperation to undergo visual function assessment (i.e. best-corrected visual acuity (BCVA), as well as the above-mentioned investigations.
4. Written, informed consent to participate in the study

Exclusion Criteria:

1. Patients with pseudo-RP
2. Patients with cystic macular lesions or progressive retinal disease due to any cause other than retinal dystrophy
3. Patients with reduced visual acuity due to media opacities (e.g. cataract).
4. Patients with any contraindication or known allergy to CAI or anti-VEGF agents
5. Patients who have undergone vitreo-retinal surgery or intravitreal injection.

Methods:

Phase 1: Patients with best corrected visual acuity (BCVA) < 0.5 will receive carbonic anhydrase inhibitors (CAI) [oral acetazolamide 500mg/day or topical brinzolamide twice daily] and followed up for three months. Baseline urea and electrolyte (U&E) will be tested prior to receiving CAI, and monitored every month while on the treatment. Upon completion of the treatment course, the patients will be assessed for response with visual function assessment and central macular thickness (CMT) on OCT. Patients who show an adequate response (defined as > 10% reduction of CMT) and/or improvement of BCVA by two lines or more) will continue in the CAI arm.

Phase 2: Patients who do not show an adequate response with CAI or develop significant side effects from CAI treatment will stop receiving CAI and will move to Phase 2 of the study and receive three 0.5mg IVR injection at monthly intervals. Upon completion of the treatment course, the patients will be assessed for response with visual function assessment and CMT on OCT.

The purpose of the proposed procedures/treatment, as well as potential complications, will be clearly explained to participants. It will be made clear to the patient that IVR treatment is experimental and may or may not lead to improvement of vision. The patient will also be informed that the treatment will be withheld in case of allergy or complications. It will be emphasized that he/she may withdraw from the study at any stage.

Patients will be under regular and close follow-up. They will be monitored for the development of any complications during the study. Any complication will be logged and treated appropriately. Patients' personal information, clinical history, examination, investigation results and progress with treatment, will be treated confidentially.

Institutional research ethics board approval will be obtained prior to the start of the study.

ELIGIBILITY:
Inclusion Criteria:

Omani patients over 18 year old, with retinal dystrophy and non-leaking macular cysts confirmed by fundus examination, electroretinography (ERG), optical coherence tomography (OCT), fundus fluorescein angiography (FFA) and genetic testing.

Included patients should also have the capacity and cooperation to undergo visual function assessment (i.e. best-corrected visual acuity (BCVA), color vision as well as the above-mentioned investigations.

Exclusion Criteria:

Patients with pseudo-retinitis pigmentosa, those with cystic macular lesions or progressive retinal disease due to any cause other than retinal dystrophy, and patients with reduced visual acuity due to media opacities (e.g. cataract). Patients with any contraindication or known allergy to brinzolamide, acetazolamide or anti-VEGF agents will not receive the respective drug, nor those who underwent intraocular surgery or injection within the last 1 month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-07-24 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2019-08-29 (Actual)

PRIMARY OUTCOMES:
Macular Cyst | 3 months
  Reduction in central macular thickness by 10%
Macula | 3 months
  Improvement in visual acuity by over one line
Complications | 3 months
  Presence of any complications from treatment

CONTACTS AND LOCATIONS:
Overall Officials: Anuradha Ganesh, MD, Study Chair — Sultan Qaboos University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moustafa GA, Moschos MM. Intravitreal aflibercept (Eylea) injection for cystoid macular edema secondary to retinitis pigmentosa - a first case report and short review of the literature. BMC Ophthalmol. 2015 Apr 30;15:44. doi: 10.1186/s12886-015-0033-z. PMID 25925748
- [Background] Artunay O, Yuzbasioglu E, Rasier R, Sengul A, Bahcecioglu H. Intravitreal ranibizumab in the treatment of cystoid macular edema associated with retinitis pigmentosa. J Ocul Pharmacol Ther. 2009 Dec;25(6):545-50. doi: 10.1089/jop.2009.0089. PMID 20028262
- [Background] Yuzbasioglu E, Artunay O, Rasier R, Sengul A, Bahcecioglu H. Intravitreal bevacizumab (Avastin) injection in retinitis pigmentosa. Curr Eye Res. 2009 Mar;34(3):231-7. doi: 10.1080/02713680802710692. PMID 19274531
- [Background] Miyata M, Oishi A, Oishi M, Hasegawa T, Ikeda HO, Tsujikawa A. Long-term efficacy and safety of anti-VEGF therapy in retinitis pigmentosa: a case report. BMC Ophthalmol. 2018 Sep 14;18(1):248. doi: 10.1186/s12886-018-0914-z. PMID 30217183